CLINICAL TRIAL: NCT03905369
Title: Focus on Values to Stimulate Shared Decisions in Patients With Thyroid Cancer: A Multifaceted COMmunication BOoster (COMBO)
Brief Title: Focus on Values to Stimulate Shared Decisions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11463
Record Dates: First submitted 2019-03-21; First posted 2019-04-05 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2022-10

CONDITIONS: Thyroid Cancer
Keywords: shared decision making; quality of life; patient-doctor communication; patient treatment preferences
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Decision Support Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision aid, SDM booster and deliberation training (Experimental): In the first arm, patients have COMBO, consisting of the decision aid, the SDM-booster, and the values deliberation training for physicians
  Interventions: Other: Decision aid and SDM booster; Other: Deliberation training
- Deliberation training (Active Comparator): In the second arm, patients have the values deliberation training for physicians alone.
  Interventions: Other: Deliberation training

INTERVENTIONS:
Other: Decision aid and SDM booster — The investigators develop the decision aid and SDM booster. The scope of the investigators of decision making combines the clinical and patient perspective. The decision aids are developed for patients with TC either newly diagnosed or patients with advanced disease, presently in the follow-up at the participating centers, covering the whole treatment trajectory of these patients (Figure 4). Three treatment decisions are considered: 1) the extent of thyroid resection, 2) the use of RAI, and 3) the initiation of TKIs.The SDM-booster is developed alongside the decision aids, as the SDM-booster (or values clarification exercise) is often a component developed together with a decision aid. The SDM-booster aims to shape patients' values regarding aspects of the decision and ensuing treatment preferences.
  Other Names: Deliberation training
  Arms: Decision aid, SDM booster and deliberation training
Other: Deliberation training — The investigators develop the deliberation training. It makes physicians more aware and responsive to patients' values. The communication training for physicians will consist of 1) an e-learning SDM-training lasting 40 minutes and, 2) an individual values deliberation training lasting 2 hours.

SUMMARY:
Most patients with non-medullary thyroid carcinoma (TC) achieve remission after primary treatment. Nonetheless, 30% develop recurrent disease and/or distant metastases resulting in worse survival. Patients with low- and intermediate-risk, whilst having a good prognosis, generally undergo similar primary treatment as those with a high-risk disease and face the risk of complications and burden of treatment, without a proven benefit in long-term outcome. For these patients, current guidelines state that less aggressive treatment (e.g. hemi-thyroidectomy vs. total thyroidectomy, and selective use of radioiodine (RAI) therapy), and tailored follow-up can be equally acceptable leaving room for patients' preferences. For high- risk patients, important unanswered question regard the optimal timing of starting tyrosine kinase inhibitors (TKI). For those who are asymptomatic or only mildly symptomatic, starting the treatment too early may expose them to side effects and impair quality of life, without evidence of a survival benefit.

Different patients have different views on these decisions, and so do physicians. Therefore, care should honour preferences and values of individual patients, and care should involve patients through shared decision making (SDM). The principle of SDM is twofold: 1. physicians provide patients with information on the existing options, and 2. help patients identify their preferences considering their individual values and needs. This involves important life values, for instance the desire to do everything possible, or to minimise complaints.

Addressing patients' treatment-related values is arguably the most difficult part of SDM so patient values are less likely to be discussed and honoured in a consultation. Current tools improve values deliberation but their effects are clearly insufficient. Tools should be integrated and applied in consultations to increase effectiveness. To strengthen values deliberation with TC as an example, a multifaceted intervention, COMBO, is proposed including 1) a patient values clarification exercise, named SDM-booster, 2) a physician values deliberation training using the SDM-booster, and 3) a patient decision aid. The SDM-booster strengthens values deliberation by 1) strengthening and clarifying patients' values and preferences, 2) communicating patients' values in the consultation, 3) serving as a focus in the values deliberation training.

ELIGIBILITY:
Decision 1: total thyroidectomy vs. hemithyroidectomy:

Inclusion Criteria:

* patients with nodules >1 cm and <4 cm, with cytology result suspicious or malignant (Bethesda 5 or 6) with no clinical or radiological evidence of pathological lymph nodes and/or distant metastases before the primary (diagnostic) surgery
* patients with histologically (after diagnostic hemithyroidectomy) proven TC but are defined as low-risk according to the ATA classification.

Exclusion criteria:

* patients with multifocal TC
* patients with incomplete resection of the primary tumor
* patients with ATA defined intermediate risk or high risk

Decision 2: no treatment with RAI vs. treatment with RAI:

Inclusion criteria:

• patients with ATA defined low-risk and patients with multifocal papillary TC in the absence of other adverse features

Exclusion criteria:

• patients with ATA defined intermediate and high risk

Decision 3: active surveillance vs. systemic treatment

Inclusion criteria:

• patients with asymptomatic or mildly symptomatic RAI-refractory (slowly) progressive metastatic disease

Exclusion criteria:

• patients with coexisting conditions that do not allow prescription of TKI's

Other exclusion Criteria:

* lack of Dutch language proficiency
* mental incompetence hampering the process of shared decision making as judged by the physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
5-item Observer OPTION scale | 2.5 years
  Audio recordings of the patient doctor communication. Measuring shared decision making by assessing recordings or transcripts of encounters from clinical settings. Each item is score 0-4 (0= no effort, 1 = minimal effort, 2 = moderate effort, 3 = skilled effort, 4 = exemplary effort), yielding a total between 0-20.

SECONDARY OUTCOMES:
Problem-Solving Decision-Making Scale from Deber | 1 year
  The problem solving decision making scale comprises six tasks, four tasks problem solving and two tasks decision making.
  All six tasks are evaluated on a 5-point Likert scale, where: 1 = the doctor alone; 2 = mostly the doctor; 3 = both equally; 4 = mostly me and 5 = me alone.
Knowledge questionnaire about treatment options | 1 year
  Objective knowledge will be measured with 5 right/wrong items about the three treatment decisions (hemithyroidectomy/total thyroidectomy, RAI/no RAI, active surveillance/TKI). These items will be generated by a panel of experts not involved in the development of the decision aid.
Decision evaluation scale | 1 year
  The Decision Evaluation Scales comprise the Satisfaction- Uncertainty, Informed Choice, and Decision Control scale. Each scale contain five items asking about the decision between screening and prohylactic mastectomy. Responses were on a 5- point scale ranging from 1 (strongly disagree) to 5 (strongly agree).
Trust in oncologist scale - short form | 1 year
  This scale assesses cancer patients' trust in their oncologist, it's a 5-item measure. Each item is scored on a five-point Likert scale: 1 = totally disagree, 2 = disagree, 3 = as much agree as disagree, 4 = agree, 5 = strongly agree
3-item Collaborate instrument | 1 year
  Patient's subjective evaluation of shared decision making process. Each item is scored 0-4 (0 = no effort was made, 1 = a little effort was made, 2 = some effort was made, 3 = a lot of effort was made, and 4 = every effort was made)

CONTACTS AND LOCATIONS:
Locations (11):
- Netherlands (11):
  - Rijnstate hospital, Arnhem, Gelderland
  - CWZ, Nijmegen, Gelderland
  - Radboudumc, Nijmegen, Gelderland
  - MUMC, Maastricht, Limburg
  - Catharina hospital, Tilburg, North Brabant
  - AUMC, Amsterdam, North Holland
  - AVL, Amsterdam, North Holland
  - LUMC, Leiden, South Holland
  - Haga, The Hague, South Holland
  - UMCG, Groningen
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No